CLINICAL TRIAL: NCT00819559
Title: Role of Preoperative Chemoradiotherapy in Clinically T3No Mid and Low Rectal Cancer : Multi-Institute Clinical Study
Brief Title: Preoperative Chemoradiotheray for Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korean Rectal Cancer Study Group (Network)
Responsible Party: Gyu-Seog Choi, Professor, School of Medicine, Kyungpook National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRCSG1
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Rectal Neoplasm
Keywords: Rectal neoplasm; Clinical stage; T3N0; Preoperative chemoradiotherapy; Laparoscopic; Open resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Open PCRT group (Active Comparator): Patients who underwent preoperative chemoradiotherapy and open resection
  Interventions: Radiation: PCRT
- Open no PCRT group (Experimental): Patients who did not undergo preoperative chemoradiotherapy and open resection
  Interventions: Radiation: PCRT
- LAP PCRT group (Active Comparator): Patients who underwent preoperative chemoradiotherapy and laparoscopic resection
  Interventions: Radiation: PCRT
- LAP no PCRT group (Experimental): Patients who did not undergo preoperative chemoradiotherapy and laparoscopic resection
  Interventions: Radiation: PCRT

INTERVENTIONS:
Radiation: PCRT — Preoperative chemoradiotherapy
  Other Names: preoperative chemoradiotherapy

SUMMARY:
Hypothesis

* Pre operative radio-chemotherapy might be not mandatory to improve local recurrent rate and survival rate in the mid-lower rectal cancer patients with T3N0 clinical stage, if surgical principals were kept.
* Laparoscopic resection is not inferior to Open surgery in the treatment of rectal cancer.

DETAILED DESCRIPTION:
It is known that 20-60% of the rectal cancer patients treated with radical resection have the local recurrence. Therefore, chemo-radiotherapy before or after operation have been the standard treatment protocol in the rectal cancer patients to reduce the local recurrence, preserve more surrounding pelvic viscera, improve the prognosis and eventually quality of life. The preoperative chemo-radiotherapy was introduced by the German Rectal Cancer study, which compared pre- and postoperative chemo and radiotherapy. In this study, the authors reported that preoperative chemo-radiotherapy reduced local recurrent rate and 3 or 4 degree toxicity and improved the compliance for treatment. Since the introduction of chemo and radiotherapy in the treatment of rectal cancer, there have been numerous controversies on the guidelines or protocols of chemo-radiotherapy. In 1990, National Institute of Health (NIH) recommended postoperative chemo- radiotherapy to all the pT3 or pN1 rectal cancer patients at the consensus conference. In some studies, they reported that good clinical outcome and low local recurrence rate were obtained by only surgical treatment in the pT3N0 rectal cancer patients with favourable pathological characteristics. They also insisted that the effectiveness of postoperative chemo- radiotherapy was not evident. Gunderson, et al. retrospectively evaluated the five-year survival rate of the pT3N0 patients. They reported that the patients with surgery and chemotherapy showed the similar survival rate with the patients who underwent surgery and postoperative chemo-radiotherapy. National Cancer Data Base showed the similar report. However, there are some problems to apply theses results to the decision of preoperative therapeutic options. Moreover, some papers showed the low local recurrent rate (less than 5%) in the stage II without the supplement therapy, when the TME was precisely performed. All these results present the controversies on the radio-chemotherapy on all the T3N0 patients in terms of the clinical outcomes and the prognosis. In Korea, numerous clinical trials have been performed on the rectal cancer patients, however there has been no clinical study for preoperative chemo- radiotherapy in the T3N0 rectal cancer patients. In this reason, the protocols are different among institutions without unified standard treatment protocol. In this study, the authors compare the accuracy of diagnosis, the functional differences according to the preoperative chemo- radiotherapy, the local recurrent rate and survival rate between the two groups of T3N0 patients; one group with preoperative chemo-radiotherapy vs. the other without. In addition, the authors evaluate the advantage of the laparoscopic surgery, such as an extensive vision, so that laparoscopy can help rectal surgery as well as the surgical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically demonstrated and cytologically evident rectal cancer (Glandular carcinoma: located on 4-12cm from anus), the case without remote metastasis
* Age: 18-70 years old
* The patients who did not undergo radiation therapy, surgery or antitumor agent therapy with the same disease medical history
* The patients with clinical stage of T3N0 identified by ultrasound or MRI
* Appropriate bone marrow, liver and renal function as follow; granulocyte ≥ 1500, platelet ≥ 80,000, bilirubin < 1.5 mg/dl , Serum Creatinine < 1.5 mg/dl, BUN < 30,
* The patients who understood the rights to withdraw the agreement at any time and signed on the informed consent form with or without their legal representatives.

Exclusion Criteria:

* Remote metastatic disease
* When the patient is concerned about the local recurrence if the preoperative chemo-radiation therapy is not undergone, or when the patient expects that the possibility of conservation of sphincter is improved owing to the preoperative chemo-radiotherapy.
* Pregnancy
* Radiotherapy, the past history of operation or chemotherapy
* Familial multiple polyp
* Uncontrolled psychiatric disorder, chronic alcohol disease or drug addiction and CNS(Central Nervous System) disorder
* Other malignant disorder
* After the radiotherapy or the case which remote metastasis is detected during the surgery
* The case which has splanchnemphraxis or the risk of progression to occlusion during the examination period
* Those patients who do not agree to participate in this study
* The patients who seemed to be likely to stop in the middle of clinical study.
* The patients who cannot undergo the regular follow-up owing to the following reasons. For instance, the patients who have psychologic, social, family or geographic reason or the patients who have difficulties in observing proper follow-up or clinical examination plan. Also, the patient who the doctor considers them as improper subjects of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-02 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 year

SECONDARY OUTCOMES:
Overall survival Local recurrence Early or late complication associated with preoperative radiotherapy Quality of life Accuracy of clinical staging Difference of surgical outcome between laparoscopic and open surgery | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gyu-Seog Choi, M.D., Principal Investigator — School of Medicine, Kyungpook National University
Locations (1):
- Korean Rectal Cancer Study Group, Daegu, South Korea